CLINICAL TRIAL: NCT02869230
Title: Radioguided Occult Lesion Localization (ROLL) is Superior a to the Wire-Guided Lesion Localization (WGLL)? Randomized Controlled Clinical Trial
Brief Title: ROLL vs WGLL for Non-palpable Breast Lesions
Acronym: ROLLvsWGLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C41030610-019
Record Dates: First submitted 2013-09-20; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Non palpable breast lesions; radioguided occult lesion localization
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radioguided occult lesion localization (Other): The ROLL technique (radioguided occult lesion localization) is characterized by the injection of a radiotracer in the center of the lesion
  Interventions: Procedure: ROLL
- wire-guided lesion localization (Experimental): wire-guided lesion localization, including better lesion centricity in relation to margins,decreased marking time, reduced surgery time, and better aesthetic outcomes
  Interventions: Procedure: wire-guided lesion localization

INTERVENTIONS:
Procedure: ROLL — The ROLL technique (radioguided occult lesion localization) is characterized by the injection of a radiotracer in the center of the lesion
  Arms: Radioguided occult lesion localization
Procedure: wire-guided lesion localization — wire-guided lesion localization, including better lesion centricity in relation to margins,decreased marking time, reduced surgery time, and better aesthetic outcomes
  Arms: wire-guided lesion localization

SUMMARY:
Here were present a controlled clinical trial comparing wire-guided lesion localization (WGLL)and radioguided occult lesion localization (ROLL) in patients treated for nonpalpable breast lesions at the Instituto Nacional de Cancerología (National Cancer Institute)in Bogotá,Colombia.

DETAILED DESCRIPTION:
The aim of this study was to compare the radioguided occult lesion localization (ROLL) technique with the wire-guided lesion localization (WGLL) technique to assess the optimal localization and excision of nonpalpable breast lesions in patients at a unique reference medical center.

A controlled clinical trial was designed to compare the WGLL and ROLL techniques in women presenting with breast lesions diagnosed by mammography or ultrasound at the Instituto Nacional de Cancerología in Bogotá, Colombia from March 2006 to June 2011.

This study evaluate 129 patients; 64 (49.6%) patients were treated using ROLL and 65 (51.4%) using WGLL.

ELIGIBILITY:
Inclusion Criteria:

* Female patients older than 18 years
* Lesions suggesting malignancy (BIRADS 4 and 5)
* Solid nodules in postmenopausal women (BIRADS 3 mammograms).

Exclusion Criteria:

* Pregnant or nursing
* Patients with suspected multifocal or multicentric disease (suspicious microcalcifications scattered over a wide area on mammography)
* Patients with retro-areola lesions (less than 2 cm away from the nipple)
* Lesions that had previously undergone surgery or excisional biopsies in the compromised breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2006-03; Primary Completion 2011-06 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Localization of nonpalpable breast lesion (percentage) | 30 days

SECONDARY OUTCOMES:
presence of malignancy | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: faustino bastidas, md, Study Chair — Instituto Nacional de Cancerologia de Mexico